CLINICAL TRIAL: NCT03878992
Title: Effects of Growth Hormone and IGF-1 on Anabolic Signals and Stem Cell Recruitment in Human Skeletal Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GHDSCs
Record Dates: First submitted 2019-03-07; First posted 2019-03-18 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-02

CONDITIONS: Growth Hormone Deficiency; Growth Hormone Treatment
Keywords: Growth hormone; Satellite cells; Metabolism; insulin-like effects
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone; Injections; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: All participants will be studies two times - one time before initiation of GH replacement therapy and one time following three months of GH replacement therapy. The two times are identical. The trial day includes infusion of tracers (glucose, tyrosine, phenylalanine, urea, palmitate), muscle biopsies, subcutaneous fat biopsies, an intravenous bolus of 0.5 mg GH, indirect calorimetry, plethysmography, blood samples, strength test, DXA scan and spectroscopy of liver and muscle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GHD (Other): GHD patients will be studied two times - one time before initiation of GH replacement therapy and one time following three months of GH replacement therapy. The two trial days are identical
  Interventions: Drug: Genotropin miniquick 0.5 mg, injection

INTERVENTIONS:
Drug: Genotropin miniquick 0.5 mg, injection — GH will be given as an injection. Muscle biopsy will be obtained from m. vests laterals of the dominant leg. Fat biopsies will be obtained from subcutaneous abdominal fat. Tracers will be given as a bolus followed by continuous infusion for 6 hours. For palmitate tracer the infusion will be for only 1,5 hours followed by a one hour break and then another 1 hour infusion. Blood tests will be drawn from a venous catheter placed on the dorsal side of the hand.
  Other Names: Muscle biopsy; fat biopsy; blood tests; pletysmography; Tracers of metabolism, infusion

SUMMARY:
12 adult hypopituitary patients with newly diagnosed Growth hormone (GH)-deficiency will be studied two times. The first examinations will be performed shortly after time of diagnose before initiation of exogenous GH treatment, where each subject will receive a single intravenous bolus of 0.5 mg GH. The examination day will be repeated after prolonged GH replacement therapy (>3 month after treatment initiation).

DETAILED DESCRIPTION:
The overarching aim of this project is to investigate the mechanisms underlying loss of muscle mass in adults (sarcopenia) and the therapeutic potential of growth hormone (GH). The underlying hypothesis is that absence of GH and subsequent reduced insulin-like growth factor I (IGF-I) will impair normal proliferation of skeletal muscle stem cells and this is associated with metabolic dysfunction.

GH is an important regulator of substrate metabolism and muscle mass. GH treatment reduces overall fat mass (FM) through lipolytic actions in adipose tissues and decreased adipose tissue triacylglycerol (TAG) synthesis. In skeletal muscle, exogenous GH administration production shifts substrate metabolism from glucose to lipid oxidation. In addition, GH mediates protein anabolic actions by production of IGF-I during sufficient nutrient supply and maintained insulin secretion. Circulating IGF-I is primarily produced in the liver, but animal studies suggest that locally produced autocrine and paracrine IGF-I is sufficient to maintain normal growth.

GH deficiency (GHD) is a rare disorder characterized by the inadequate secretion of GH from the anterior pituitary gland and requires treatment with exogenous GH administration. Cell culture studies demonstrates that GH elicits insulin-like effects in cells deprived of GH. GH exerts its biological effects through binding to site 1 and 2 on the extracellular domain of a preformed GHR dimer. GHR activation initiates auto-phosphorylation of the receptor-associated Janus Kinase 2 (JAK2), which subsequently induces GHR cross-phosphorylation. The insulin-like effects are mediated by tyrosine phosphorylation of downstream targets including insulin receptor substrate-1 (IRS-1) and IRS-2. During physiological conditions, this signaling pathway is inhibited by the actions of a class of proteins known as suppressors of cytokine signaling (SOCSs).

GHD in adults can be acquired as a result of trauma, infection, radiation therapy, or tumor growth within the brain. It is characterized by a number of variable symptoms including reduced energy levels, altered body composition and reduced muscle strength. Satellite cells (SCs), the skeletal muscle stem cells, are essential for muscle regeneration in genetic or autoimmune muscle diseases as well as after ischemic, chemical or mechanical trauma to the myofibers. Furthermore, SCs are the primary source to supply new myonuclei to growing myofibers during non-traumatic mechanical overload. In rats, GH-administration increases number of SCs in cross-sections of muscle fibres22, and fibre type composition in skeletal muscle is altered in animals with GHD. Together these findings indicate an importance of GH and IGF-I stimulation for muscle regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed adult onset growth hormone deficiency

Exclusion Criteria:

* Documentation of Growth hormone deficiency for less than three months
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Phosphorylation of Akt in muscle biopsies | Analyses will be performed through study completion, an expected average of 1.5 years
  Muscle biopsies will be analysed for phosphorylation of Akt

SECONDARY OUTCOMES:
Satellite cell count | Analyses will be performed through study completion, an expected average of 1.5 year
  The number of Satellite cells per muscle fiber will be analysed on muscle cross sections from muscle biopsies
Satellite cell proliferation and differentiation in cell culture | Analyses will be performed through study completion, an expected average of 1.5 year
  Analyses of satellite cells ability to proliferate and differentiate will be performed on cell culture following fluorescent activated cell sorting. Comparison will be between first and second visit.
Strength of muscle | Analyses will be performed through study completion, an expected average of 1.5 year
  assessed by isokinetic/dynamic measurements using a dynamometer
Muscle mass | Analyses will be performed through study completion, an expected average of 1.5 year
  Qualified by DXA scan
Glucose turnover rate | Analyses will be performed through study completion, an expected average of 1.5 year
  Evaluated through blood samples
Fatty acid turn over rate | Analyses will be performed through study completion, an expected average of 1.5 year
  evaluated through blood samples
Urea turnover rate | Analyses will be performed through study completion, an expected average of 1.5 year
  evaluated by blood samples and urin collection

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto Jørgensen, Professor, Study Chair — Aarhus University Hospital
Locations (1):
- Department of Endcrinology, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
There is no specific plan to share IPD at the moment. If this should be of interest it will only happen after approval from the local ethics committee

REFERENCES:
- [Background] Zurlo F, Larson K, Bogardus C, Ravussin E. Skeletal muscle metabolism is a major determinant of resting energy expenditure. J Clin Invest. 1990 Nov;86(5):1423-7. doi: 10.1172/JCI114857. PMID 2243122
- [Background] DeFronzo RA, Jacot E, Jequier E, Maeder E, Wahren J, Felber JP. The effect of insulin on the disposal of intravenous glucose. Results from indirect calorimetry and hepatic and femoral venous catheterization. Diabetes. 1981 Dec;30(12):1000-7. doi: 10.2337/diab.30.12.1000. No abstract available. PMID 7030826
- [Background] Nellemann B, Vendelbo MH, Nielsen TS, Bak AM, Hogild M, Pedersen SB, Bienso RS, Pilegaard H, Moller N, Jessen N, Jorgensen JO. Growth hormone-induced insulin resistance in human subjects involves reduced pyruvate dehydrogenase activity. Acta Physiol (Oxf). 2014 Feb;210(2):392-402. doi: 10.1111/apha.12183. Epub 2013 Nov 22. PMID 24148194
- [Background] Salomon F, Cuneo RC, Hesp R, Sonksen PH. The effects of treatment with recombinant human growth hormone on body composition and metabolism in adults with growth hormone deficiency. N Engl J Med. 1989 Dec 28;321(26):1797-803. doi: 10.1056/NEJM198912283212605. PMID 2687691
- [Background] Rosenbaum M, Gertner JM, Leibel RL. Effects of systemic growth hormone (GH) administration on regional adipose tissue distribution and metabolism in GH-deficient children. J Clin Endocrinol Metab. 1989 Dec;69(6):1274-81. doi: 10.1210/jcem-69-6-1274. PMID 2685009
- [Background] Pochini L, Oppedisano F, Indiveri C. Reconstitution into liposomes and functional characterization of the carnitine transporter from renal cell plasma membrane. Biochim Biophys Acta. 2004 Feb 10;1661(1):78-86. doi: 10.1016/j.bbamem.2003.12.001. PMID 14967477
- [Background] Ridderstrale M. Signaling mechanism for the insulin-like effects of growth hormone--another example of a classical hormonal negative feedback loop. Curr Drug Targets Immune Endocr Metabol Disord. 2005 Mar;5(1):79-92. doi: 10.2174/1568008053174787. PMID 15777207
- [Background] Vahl N, Jorgensen JO, Jurik AG, Christiansen JS. Abdominal adiposity and physical fitness are major determinants of the age associated decline in stimulated GH secretion in healthy adults. J Clin Endocrinol Metab. 1996 Jun;81(6):2209-15. doi: 10.1210/jcem.81.6.8964853.
- [Background] Vahl N, Jorgensen JO, Skjaerbaek C, Veldhuis JD, Orskov H, Christiansen JS. Abdominal adiposity rather than age and sex predicts mass and regularity of GH secretion in healthy adults. Am J Physiol. 1997 Jun;272(6 Pt 1):E1108-16. doi: 10.1152/ajpendo.1997.272.6.E1108. PMID 9227458
- [Background] Rasmussen MH, Hvidberg A, Juul A, Main KM, Gotfredsen A, Skakkebaek NE, Hilsted J, Skakkebae NE. Massive weight loss restores 24-hour growth hormone release profiles and serum insulin-like growth factor-I levels in obese subjects. J Clin Endocrinol Metab. 1995 Apr;80(4):1407-15. doi: 10.1210/jcem.80.4.7536210.
- [Background] Meinhardt UJ, Ho KK. Modulation of growth hormone action by sex steroids. Clin Endocrinol (Oxf). 2006 Oct;65(4):413-22. doi: 10.1111/j.1365-2265.2006.02676.x. PMID 16984231
- [Background] Ullman M, Oldfors A. Effects of growth hormone on skeletal muscle. I. Studies on normal adult rats. Acta Physiol Scand. 1989 Apr;135(4):531-6. doi: 10.1111/j.1748-1716.1989.tb08612.x. PMID 2735197